CLINICAL TRIAL: NCT05051605
Title: Evaluation of the Immune Response to COVID-19 Vaccine in Recipients of Living Donor Liver Transplantation
Brief Title: Immune Response to COVID-19 Vaccine in Recipients of Living Donor Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Sayed Fouad, Principal investigator, Ain Shams University
Other Study IDs: RHDIRB2020110301 REC 45
Record Dates: First submitted 2021-09-17; First posted 2021-09-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Liver Transplant
Keywords: Liver; transplantation; COVID-19; Coronavirus; Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinated group: Fifty living donor liver transplantation recipients on maintenance immunosuppressive regimen who would receive COVID-19 vaccine at least 3 months postoperatively.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Severe acute respiratory syndrome- coronavirus-2 (SARS-CoV-2)vaccine according to vaccine availability in the Egyptian ministry of health.

SUMMARY:
A prospective cohort study to evaluate the response to COVID-19 vaccine in liver transplantation patients.

DETAILED DESCRIPTION:
fifty living donor liver transplantation recipients during maintenance immunosuppression phase will be vaccinated against COVID-19 followed by assessment of immune response to the vaccine and further investigation of correlation of immune response to genetic polymorphisms of HLA DRB1(rs2647087) gene and IL-18 (rs187238 and rs917997) gene.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* At least 3 month post transplantation

Exclusion Criteria:

* pediatric recipients
* Active covid infection at the time of the study
* Pregnancy
* Allergy to any ingredients included in the vaccine
* Lactation in first six month of delivery
* Active Acute cellular rejection proven by liver biopsy
* Acute Febrile state with either leucopenia or leucocytosis
* High dose of corticosteroid at study timing (pulse methyl prednisolone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living donor liver transplantation recipients willing to be vaccinated against COVID-19 and capable of signing an informed consent to participate in this cohort
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody titer change 14 days after vaccination compared to baseline | At baseline, at 14 days after whole course of vaccination
  neutralizing antibody response to SARS-CoV-2 vaccine in recipients post living donor liver transplantation
Neutralizing antibody titer change 28 days post vaccination compared to baseline | At baseline and 28 days after whole course of vaccination
  neutralizing antibody response to SARS-CoV-2 vaccine in recipients post living donor liver transplantation

SECONDARY OUTCOMES:
Interleukin-6 serum level | At baseline, at 14 and 28 days after whole course of vaccination
  Assessing the cellular immunological response to SARS-CoV-2 vaccine in recipients post living donor liver transplantation
Incidence of confirmed coronavirus disease | 28 days after whole course of vaccination
  Patient follow-up for confirmed symptomatic infection by SARS-COV2 virus
Incidence of adverse events related to vaccine | 7 days after each dose of the vaccine and up to 28 days after last vaccine dose administered
  Self reported safety and tolerability of vaccine
Incidence of acute graft rejection | On 14 and 28 days post whole course vaccination
  Follow-up for signs and symptoms of graft rejection
Immune response correlation to HLA DRB1 genetic polymorphism | 28 days post whole course vaccination
  TaqMan®️ SNP genotyping assay of HLA DRB1 gene (rs2647087)
Immune response correlation to IL-18 genetic polymorphism | 28 days post whole course vaccination
  TaqMan®️ SNP genotyping assay of IL-18 gene (rs187238 and rs917997)

CONTACTS AND LOCATIONS:
Overall Officials: Rana Sayed, PhD, Study Director — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain Shams center for organ transplantation (ASCOT), Ain shams university specialized hospital, Cairo, Please Select Region, State Or Province, Egypt